CLINICAL TRIAL: NCT05270083
Title: Role of NeuraceqTM (Florbetaben F18 Injection) PET in Young Athletes With and Without Persistent Cognitive Complaints Following Multiple Concussions: A Pilot Study
Brief Title: Neuraceq™ PET for Detection of Brain Changes in Young Athletes Post-concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Marc A. Seltzer, Principal Investigator, Section Chief, Diagnostic Radiology, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D16096
Record Dates: First submitted 2022-02-24; First posted 2022-03-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Athletes with mild to moderate traumatic brain injury (mTBI) and good outcome (Active Comparator): Young athletes who have sustained one or more concussions without persistent cognitive complaints at least one year post-injury
  Interventions: Diagnostic Test: NeuraCeq PET imaging with intravenous (IV) dose of 300MBq of Neuraceq™ ([F-18]Florbetaben)
- Athletes with persistent cognitive deficits due to mild to moderate traumatic brain injury (mTBI) (Active Comparator): Young athletes who have sustained one or more concussions with persistent cognitive complaints at least one year post-injury in spite of medical and cognitive treatment intervention.
  Interventions: Diagnostic Test: NeuraCeq PET imaging with intravenous (IV) dose of 300MBq of Neuraceq™ ([F-18]Florbetaben)

INTERVENTIONS:
Diagnostic Test: NeuraCeq PET imaging with intravenous (IV) dose of 300MBq of Neuraceq™ ([F-18]Florbetaben) — Participants will receive an intravenous (IV) dose of 300 MBq of Neuraceq™ in a volume of 10 mL or less. A 30 minute duration PET image will be acquired starting immediately after Neuraceq™ injection. A second 20-minute duration PET image will be acquired starting 90 minutes after Neuraceq™ injection.
  Other Names: 18F-Florbetaben

SUMMARY:
The purpose of the study is to learn if Neuraceq™ (Florbetaben F 18 Injection) PET can detect changes in the brains of young athletes who sustained one or more concussions with or without persistent cognitive complaints at least 5 years after injury.

DETAILED DESCRIPTION:
Former college athletes who sustained at least one previous concussion will undergo computerized neurocognitive testing and a structured questionnaire of present symptoms. [F-18] Florbetaben PET images will be acquired dynamically, with data binned in 20 time frames of 1 min each (early phase), followed by 4 frames of 5 min each (late phase), with image frames summed within each phase after linearly coregistering to subjects' mean images, then elastically transformed to template space of a florbetaben scan used in standardized volume of interest quantification, and intensity normalized to mean voxel value within each phase.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* A minimum of 1 concussion prior to study entry
* A minimum of one year post first concussion
* mTBI as defined by the American Congress of Rehabilitative Medicine
* Participants in Cohort A must have either subjective or objective evidence of persistent cognitive deficits

Exclusion Criteria:

* Impaired decision-making capacity, i.e. inability to provide informed consent
* Pregnancy
* History of other neurologic disorders (e.g., epilepsy, cerebrovascular disease, neurodegenerative disorders, intellectual disability)
* Significant systemic medical illness
* Current DSM-IV Axis I diagnosis of psychiatric illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Neuraceq™ PET Imaging | Up to 90 minutes after injection
  Participants will receive an intravenous (IV) dose of 300 MBq of Neuraceq™ ([F-18]Florbetaben) in a volume of 10 mL or less. A 30 minute duration PET image will be acquired starting immediately after Neuraceq™ injection. A second 20-minute duration PET image will be acquired starting 90 minutes after Neuraceq™ injection. Imaging data will be reconstructed using standard iterative reconstruction algorithm and with CT-based attenuation correction. Images will be interpreted both visually and semi-quantitatively (cortical-to-cerebellum standardized uptake value rations) for 6 target cortical regions of interest (frontal, temporal, parietal, anterior cingulate, posterior cingulate, and precuneus), using the whole cerebellum as the reference region.
Cognitive Assessment_1 | within 24 hours of [F-18]Florbetaben PET imaging
  Participants will complete a set of cognitive questionnaires to assess presence or absence of cognitive complaints. Altered cognitive performance will be defined as either one score of more than 2 standard deviations or two scores of 1 standard deviation below the age-adjusted norm or estimates of baseline premorbid function (using the Barona Index) on tests of attention and/or memory.
Cognitive Assessment_2 | within 24 hours of [F-18]Florbetaben PET imaging
  Participants will complete a set of cognitive questionnaires to assess presence or absence of cognitive complaints. Significant cognitive complaints will be defined as scores of 1 standard deviation below the mean on the Multiple Ability Self-Report Questionnaire (MASQ).

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Seltzer, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No